CLINICAL TRIAL: NCT05342337
Title: Investigation of the Effectiveness of Biopsychosocial Exercise Therapy Approach With Telerehabilitation in Patients Living With HIV
Brief Title: Exercise Therapy With Telerehabilitation in Patients Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aysenur Tuncer, Assistant Professor, Hasan Kalyoncu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/024
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections
Keywords: HIV; Telerehabilitation; Biopsychosocial Approach
MeSH Terms: conditions — HIV Infections | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): The Telerehabilitation program includes a Biopsychosocial Exercise Therapy (BETY) approach.
  BETY approach includes patient education on pain, functional body stabilization exercises (mind-body information management), dance therapy authentic movement (emotion-state information management), and sexual information management.
  Interventions: Other: Telerehabilitation Group
- Control Group (Active Comparator): The control group participants include those who do not want to receive exercise treatment with telerehabilitation and take their routine medications during the 12 weeks period.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Telerehabilitation Group — The Telerehabilitation program includes a Biopsychosocial Exercise Therapy (BETY) approach.
  BETY approach includes patient education on pain, functional body stabilization exercises (mind-body information management), dance therapy authentic movement (emotion-state information management), and sexual information management.
  Telerehabilitation group participate in the sessions that last for one and a half hours, 3 days a week for 12 weeks, video conference over the Zoom program. The investigator, who provides supervision during the sessions, also participates in the exercises simultaneously.
  Arms: Telerehabilitation Group
Other: Control group — The control group participants include those who do not want to receive exercise treatment with telerehabilitation and take their routine medications during the 12 weeks period.
  Arms: Control Group

SUMMARY:
To investigate the effectiveness of the Biopsychosocial Exercise Therapy Approach (BETY) approach with the Telerehabilitation in patients living with HIV (PLWH).

DETAILED DESCRIPTION:
55 individuals living with HIV (PLWH) were included in the study. Among those individuals, 25 individuals who volunteer to exercise with telerehabilitation will be grouped in the telerehabilitation group. The rest of the individuals who do not participate in the exercise group will be in the control group.

Group 1: Telerehabilitation group: Individuals in the telerehabilitation group attend sessions that last for one and a half hours, 3 days a week for 12 weeks, in the company of an investigator over the videoconference through zoom. The investigator, who provides supervision during the sessions, also participates in the exercises simultaneously.

Group 2: Control group: Individuals in the control group continue their routine drugs.

Both the telerehabilitation exercise group and the control group continue their drug treatments during the 12 weeks of the period.

ELIGIBILITY:
Inclusion Criteria:

* Patients living with HIV (PLWH),
* Ages between 18 and 65 years old,
* Participants attend and follow instructions through telerehabilitation.

Exclusion Criteria:

* Participants who use recreational drugs
* Participants who do not adapt to the exercises through telerehabilitation,
* Participants who did not agree to be volunteers are not included in our study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Biopsychosocial Exercise Therapy Questionnaire (BETY-BQ) at 12 weeks | Baseline, 12 weeks
  The Biopsychosocial Exercise Therapy Questionnaire (BETY-BQ), consists of 30 questions. Each of the items on the scale is scored between 0-and 4 in accordance with the Likert system. A higher score indicates a poor biopsychosocial status (4: Yes always, 3: Yes often, 2: Yes sometimes, 1: Yes rarely, 0: No, never).
Change from Baseline in Short Form-36 (SF-36) at 12 weeks | Baseline, 12 weeks
  The Short Form-36 (SF-36) scale, is the most commonly used quality of life scale that evaluate physical and mental health. İt consists of 8 subscales. These subscales, physical function, physical orientation role restriction, pain, general health, vitalization, social function, emotional role restrictiveness, and mental health. Points range from 0-to 100 and the best health status of 100 points shows the worst health status of 0 points.
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) at 12 weeks | Baseline, 12 weeks
  The HADS is a self-rating scale. It contains two subscales measuring symptoms of depression (HADS-D) and anxiety (HADS-A) during the previous week. It includes seven statements on each disorder, and each response consists of a four-point rating scale (0 to 3); a higher score depicts a worse condition. For each subscale, the total score is at most 21. A score of ≥11 is considered a clinically significant disorder, whereas a score between 8 and 10 suggests a mild disorder.
Change from Baseline in FRAIL scale at 12 weeks | Baseline, 12 weeks
  The FRAIL scale is a clinical frailty screening tool. It consists of five components: Fatigue, resistance, ambulation, illness, and loss of weight (score range 0-5), and evaluates the status and severity of frailty. The presence of ≥3 components in a participants is considered frailty, while the presence of more components indicates more serious vulnerability.
Change from Baseline in Clinical Frailty Scale (CFS) scale at 12 weeks | Baseline, 12 weeks
  The Clinical Frailty Scale is an inclusive 9-point scale to summarize the overall level of fitness or frailty of participants. The scale can be easily applied to the participants. İt is based on a subjective clinical assessment categorized by the investigators. A clinical fragile scale score greater than four is to be fragility and clinical indicator. Higher scores mean greater risk.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No